CLINICAL TRIAL: NCT03269253
Title: Maternal Loss of Control Eating: a Longitudinal Study of Maternal and Child Outcomes
Brief Title: Maternal Loss of Control Eating
Status: Completed | Type: Observational
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Sponsor
Other Study IDs: GCO 15-1668
Record Dates: First submitted 2017-08-29; First posted 2017-08-31 (Actual); Last update posted 2017-08-31 (Actual); Status verified 2017-08

CONDITIONS: Eating Disorder; Obesity
Keywords: ALSPAC; longitudinal
MeSH Terms: conditions — Feeding and Eating Disorders; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study focused on investigating the effects of maternal disordered eating on maternal and child outcomes as part of a secondary data analysis of the Avon Longitudinal Study of Parents and Children (ALSPAC).

DETAILED DESCRIPTION:
Deidentified and anonymised data already collected as part of the ALSPAC study will be analysed to investigate the effects of maternal eating on maternal and child outcomes (diet, eating, weight, metabolic). The Avon Longitudinal Study of Parents and Children (ALSPAC) is a longitudinal, prospective study designed to examine the effects of environment, genetics and other factors on health and development.All pregnant women living in the geographical area of Avon, UK, who were expected to deliver their baby between 1st April 1991 and 31st December 1992, were recruited. 14,541 women were enrolled. Amongst these pregnancies, there were a total of 14,676 fetuses, resulting in 14,062 live births and 13,798 children who were alive at 1 year of age and were singletons. The ALSPAC study website contains details of all the data that is available through a fully searchable data Dictionary (http://www.bris.ac.uk/alspac/researchers/data-access/data-dictionary/).

Missingness will be assessed and standard data analytical techniques such as MI will be used.Crude and adjusted logistic, linear, and multinomial regression models will be employed.

ELIGIBILITY:
Inclusion Criteria:

-

Exclusion Criteria:

* multiple pregnancies
* no questionnaire data at 32 weeks.

eligibility criteria : enrolled in the ALSPAC study; inclusion: all women part of the ALSPAC study;

Ages: 16 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes
Study Population: All pregnant women living in the geographical area of Avon, UK, who were expected to deliver their baby between 1st April 1991 and 31st December 1992, were recruited. 14,541 women were enrolled. Amongst these pregnancies, there were a total of 14,676 fetuses, resulting in 14,062 live births and 13,798 children who were alive at 1 year of age and were singletons.
Sampling Method: Non-Probability Sample
Enrollment: 14451 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-07-20 (Actual); Study Completion 2017-07-20 (Actual)

PRIMARY OUTCOMES:
birth weight | Day 1
  weight at birth

SECONDARY OUTCOMES:
BMI | average 21 years
  body mass index
Food Frequency Questionnaire (FFQ) | average 9 months
  adult dietary patterns - software specific to the FFQ will be used to analyze data.
Food Frequency Questionnaire | average 21 years
  child dietary patterns- software specific to the FFQ will be used to analyze data.

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Micali, MD, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Micali N, Al Essimii H, Field AE, Treasure J. Pregnancy loss of control over eating: a longitudinal study of maternal and child outcomes. Am J Clin Nutr. 2018 Jul 1;108(1):101-107. doi: 10.1093/ajcn/nqy040. PMID 29873682